CLINICAL TRIAL: NCT03645187
Title: Evaluation of Anticancer Effect of Celecoxib as Adjuvant Therapy to Chemotherapy in Patients With Metastatic Colorectal Cancer
Brief Title: Celecoxib as Adjuvant Therapy to Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: celecoxib
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Colon Cancer Stage
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFERI (Active Comparator): FOLFERI regien
  Interventions: Drug: FOLFERI
- FOLFERI and celecoxib (Active Comparator): FOLFERI and celecoxib
  Interventions: Drug: Folferi and celecoxib

INTERVENTIONS:
Drug: FOLFERI — FOLFERI regimen
  Arms: FOLFERI
Drug: Folferi and celecoxib — Folferi regimen and celecoxib
  Arms: FOLFERI and celecoxib

SUMMARY:
The study aimed at evaluation of anticancer effect of celecoxib as adjuvant therapy to chemotherapy in patients with metastatic colorectal cancer

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate the anticancer effect of celecoxib as adjuvant therapy to chemotherapy in patients with metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* advanced colorectal cancer

Exclusion Criteria:

* cerebral metastases
* other malignancy
* H pylori infection
* thromboembolism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with improved radiology | 6 months
  number of patients with improved radiology

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M Mostafa, Prof, Principal Investigator — Clinical pharmacy Department- Tanta University; Mohamed Alm El-din, prof, Study Director — Clinical Oncology - Tanta University; Amira Roushdy, Msc, Study Director — Clinical pharmacy Department- Tanta University
Locations (1):
- Amira Roushdy, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mostafa TM, Alm El-Din MA, Rashdan AR. Celecoxib as an adjuvant to chemotherapy for patients with metastatic colorectal cancer: A randomized controlled clinical study. Saudi Med J. 2022 Jan;43(1):37-44. doi: 10.15537/smj.2022.43.1.20210574. PMID 35022282